CLINICAL TRIAL: NCT03135938
Title: Grading Versus Classic Inferior Oblique Anterior Transposition in Patient With Asymmetric Dissociated Vertical Deviation
Acronym: Grading vs
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Ophthalmic Research center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 95100
Record Dates: First submitted 2017-04-20; First posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Asymmetric Dissociated Vertical Deviation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grading Inferior Oblique Anterior Transposition (Active Comparator): in the classic group, IO muscle will be sutured to the sclera at the level of inferior rectus (IR) insertion at its temporal border, without considering the asymmetric DVD between the two eyes
  Interventions: Procedure: Grading Inferior Oblique Anterior Transposition surgery
- Classic Inferior Oblique Anterior Transposition (Active Comparator): in the grading group, IO muscle of the eye with more severe DVD will be sutured at the level of IR insertion and IO muscle of the eye with lower magnitude of DVD will be sutured 2mm posterior to the sclera to consider the preoperative DVD difference between the two eyes
  Interventions: Procedure: Classic Inferior Oblique Anterior Transposition surgery

INTERVENTIONS:
Procedure: Grading Inferior Oblique Anterior Transposition surgery — in the grading group, IO muscle of the eye with more severe DVD will be sutured at the level of IR insertion and IO muscle of the eye with lower magnitude of DVD will be sutured 2mm posterior to the sclera to consider the preoperative DVD difference between the two eyes.
  Arms: Grading Inferior Oblique Anterior Transposition
Procedure: Classic Inferior Oblique Anterior Transposition surgery — in the classic group, IO muscle will be sutured to the sclera at the level of inferior rectus (IR) insertion at its temporal border, without considering the asymmetric DVD between the two eyes
  Arms: Classic Inferior Oblique Anterior Transposition

SUMMARY:
Purpose: To determine the surgical outcomes of the grading versus classic Inferior Oblique Anterior Transposition (IOAT) technique in treatment of patients with asymmetric dissociated vertical deviation (DVD) and inferior oblique overaction (IOOA).

Methods: In this randomized clinical trial, a total of 38 patients with IOOA of >+1 and a minimum DVD difference of 5pd between their two eyes will be included. Comprehensive ophthalmic examinations including visual acuity assessment, measurements of noncyclo- and cycloplegic refraction as well as ocular deviation, biomicroscopic and funduscopic evaluation will be performed at baseline and repeated three months after the surgery. The function of extra ocular muscles will be evaluated by duction and version movements denoting from -4 (underaction) to +4 (overaction) grades. Also, IOOA will be graded as +1 to +4 according to the covering of the cornea under the superior eyelid during the ocular movement towards supra-nasal direction. The difference of DVD≥5pd between two eyes will be considered as asymmetric DVD. All patients will be randomized in the two groups to undergo IOAT surgical procedure; in the classic group, IO muscle will be sutured to the sclera at the level of inferior rectus (IR) insertion at its temporal border, without considering the asymmetric DVD between the two eyes; while in the grading group, IO muscle of the eye with more severe DVD will be sutured at the level of IR insertion and IO muscle of the eye with lower magnitude of DVD will be sutured 2mm posterior to the sclera to consider the preoperative DVD difference between the two eyes.

ELIGIBILITY:
Inclusion Criteria:

- Overaction of inferior oblique muscle ≥+1 and asymmetric dissociated vertical deviation >5pd between their two eyes.

Exclusion Criteria:

* Mental retardation
* Nystagmus
* Cerebral palsy
* History of ptosis and previous surgery on any cyclovertical muscle
* Restrictive or paralytic ocular deviations
* Inability to maintain fixation by each eye
* Best corrected visual acuity <20/200
* Ocular and/or systemic anomalies
* Follow up less than three months

Ages: 7 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 38 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2017-11-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference of DVD between two eyes | three months after the surgery
  alternative prism cover test

SECONDARY OUTCOMES:
Inferior oblique overaction | three months after the surgery
  Evaluation of ocular motility in 9 visual gazes

CONTACTS AND LOCATIONS:
Locations (1):
- Islamic Republic of Iran, Tehrān, Iran